CLINICAL TRIAL: NCT01339338
Title: Comparison of the Warm and Cold Contrast Media for Hysterosalpingography: a Prospective, Randomized Study
Brief Title: Warming Contrast Media for Hysterosalpingography
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: YiYang Zhu/Centra for Reproductive Medicine, Taizhou hospital of Zhejiang Province
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Taizhou200935
Record Dates: First submitted 2011-04-12; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- warm media (Experimental): Subjects undergo HSG using a warm media heated with a 37℃ water-bathing
  Interventions: Procedure: warming the contrast media
- cold media (No Intervention): the contrast media under room temperature without heat
  Interventions: Procedure: warming the contrast media

INTERVENTIONS:
Procedure: warming the contrast media — warm the contrast media with 37℃ water-bathing
  Other Names: warm media

SUMMARY:
The purpose of this study is to compare the use of warm-media with cold-media in performing hysterosalpingography (HSG).

DETAILED DESCRIPTION:
As an essential step of the infertile work-up, hysterosalpingography remains widely used in many country since it was first reported at 1914. Although HSG is a non-invasive and safety procedure, it still has some adverse. Lower abdominal pain and vasovagal episodes are mainly acute reactions to the contrast media of HSG, the later include nausea, Vomit, Sweating, Weakness and even bradycardia, occur in 16-54% of patients undergoing HSG.

Many techniques were developed to reduce adverse reactions or alleviate the pain in using of contrast media, include previous analgesia, pretreatment with corticosteroids and using non-ionic contrast media for HSG. However, in a recently Cochrane's review, reported it lack of benefit for using any pain relief medication in HSG.

Pre-Warming the hands and instruments makes physical examination more comfortable for the patients. Local active warming can valid lessen the acute pelvic pain. Experiences from the peritoneal dialysis and the laparoscopy surgical reveal that warm dialysis solution or air insufflation can decrease the pain of operation. A randomize study on Sonohysterography (SHG), another technique for exam tubal and uterine cavity diseases, cue that warming of Echovist contrast media to body temperature is a simple and effective intervention in reducing discomfort at the time exam.Because the less volume of medium injected during the HSG and the iodine medias may have different properties to the Echovist media, whether this intervention is also valid in HSG remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* infertile women who seeking for HSG testing

Exclusion Criteria:

* suspect of pregnancy
* acute low reproductive duct infection
* a known hypersensitivity to iodine
* genital bleeding
* genital malignancy

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
incidence of vasovagal episodes | from the injection of the media to a half hour after HSG
  vasovagal episodes include nausea, Vomit, Sweating, Weakness and bradycardia occurred in HSG

SECONDARY OUTCOMES:
Visual analogue scale pain score during HSG | within the first 30 seconds after the constra media "spill out"
  assessing the average pain score during HSG,Immediately after the constra media "spill out" the tubal fimbria and spread into periotneum.
Visual analogue scale pain score after HSG | a half hour after HSG
  10cm Visual analogue scale pain score after HSG

CONTACTS AND LOCATIONS:
Overall Officials: YiYang Zhu, MD, Study Director — Centra for Reproductive Medicine of Taizhou hospital
Locations (1):
- Taizhou Hospital of zhejiang Province, Taizhou, Zhejiang, China

REFERENCES:
- [Derived] Zhu YY, Mao YZ, Wu WL. Comparison of warm and cold contrast media for hysterosalpingography: a prospective, randomized study. Fertil Steril. 2012 Jun;97(6):1405-9. doi: 10.1016/j.fertnstert.2012.02.039. Epub 2012 Mar 27. PMID 22459631